CLINICAL TRIAL: NCT03486353
Title: A Phase 2 Study of FF-10501-01 in Combination with Azacitidine in Patients with Myelodysplastic Syndrome
Brief Title: A Study of FF-10501-01 in Combination with Azacitidine in Patients with Myelodysplastic Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Program terminated
Sponsor: Fujifilm Pharmaceuticals U.S.A., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FF1050101US201
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2021-07

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: myelodysplastic syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Intervention Model Description: open-label, Simon 2-stage clinical study of the combination of FF-10501-01 and azacitidine in MDS patients. The Phase 2 portion of the trial will be preceded by a Phase 1 "run-in" to evaluate the safety of the combination of FF-10501-01 plus azacitidine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Run-In Phase, Regimen 1 (Experimental): Patients will be treated with FF-10501-01 at a dose of 400 mg/m2 twice daily (BID) for 14 days plus azacitidine at a dose of 75 mg/m2 either subcutaneously (SC) or intravenously (IV) x 7 days every 28 days. One treatment cycle will be 28 days in duration.
  Interventions: Drug: FF-10501-01; Drug: Azacitidine
- Run-In Phase, Regimen 2 (Experimental): Patients will be treated with FF-10501-01 at a dose of 400 mg/m2 BID for 21 days plus azacitidine at a dose of 75 mg/m2 either SC or IV x 7 days every 28 days.
  Interventions: Drug: FF-10501-01; Drug: Azacitidine

INTERVENTIONS:
Drug: FF-10501-01 — FF-10501-01 round film-coated tablets are immediate release and come in 3 dosage strengths: 50 mg (tan), 100 mg tablets (red) and 200 mg (yellow). Each tablet contains the active ingredient (FF-10501-01 white crystalline powder) and other excipients. All dosage strengths are packaged 32 tablets to a bottle. FF-10501-01 should be stored at room temperature (20 - 25 °C).
Drug: Azacitidine — azacitidine at a dose of 75 mg/m2 either subcutaneously (SC) or intravenously (IV) x 7 days every 28 days

SUMMARY:
The primary objective of the study is to determine the response rate according to the International Working Group Response criteria for the combination of FF-10501-01 and azacitidine in patients previously untreated with hypomethylating agents, with Int2/High risk MDS according to the IPSS, and Intermediate/High/Very-High risk MDS according to the IPSS-R, or who are otherwise candidates for treatment with azacitidine.

DETAILED DESCRIPTION:
This is an open-label, Simon 2-stage clinical study of the combination of FF-10501-01 and azacitidine in previously untreated patients with high-risk MDS, or in patients with myelodysplastic syndrome (MDS) who are otherwise candidates for treatment with azacitidine in the judgment of the Investigator. The Phase 2 portion of the trial will be preceded by a Phase 1 "run-in" to evaluate the safety of the combination of FF-10501-01 plus azacitidine.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age
2. MDS as determined by bone marrow aspirate and/or biopsy according to the WHO Classification within 6 weeks of the first dose of study medication, with bone marrow blast counts of < 20%.
3. Int2/High-risk MDS according to the IPSS, Intermediate/high/very high-risk MDS according to the IPSS-R, or otherwise eligible for treatment with azacitidine in the judgment of the Investigator
4. ECOG Performance Score of 0 or 1
5. Adequate hepatic function as evidenced by AST/ALT < 3X the ULN and total bilirubin < 2X the ULN for the reference lab
6. Adequate renal function as evidenced by serum creatinine < 2 mg/dL or a calculated creatinine clearance of > 50 mL/min

Exclusion Criteria:

1. A current infection requiring treatment with intravenous antibiotics, anti-fungal agents, or anti-viral agents
2. Previous treatment with a hypomethylating agent, an HDAC inhibitor, or any other drug intended for the treatment of MDS other than hematopoietic growth factors, immunosuppressive therapy or hydroxyurea. Patients with 5q deletions may have received prior lenalidomide.
3. Use of hematopoietic growth factors (erythropoietin, G-CSF, GM-CSF, thrombopoietin receptor agonists) or immunosuppressive treatments within 7 days of first dose of study medication
4. Administration of any investigational agent within 5 half-lives of the agent; if the half-life is not known, use of such an agent within 2 weeks of the first dose of study medication
5. Active infection with HIV or hepatitis B or C; patients with a history of such disorders should undergo serological testing to evaluate the activity of the infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Response Rate | 24 months
  The primary efficacy assessment will be the objective response rate, composed of those patients who achieve a best response of CR, mCR, PR or HI based on the Modified IWG Response Criteria in MDS

SECONDARY OUTCOMES:
Hematologic Improvement Rate | 24 months
  Determination of the hematologic improvement rate for erythroid, platelet and/or neutrophil response. The number of patients who achieve trilineage hematologic improvement will be reported, as will the number who achieve improvement in each of the cell series (i.e., erythroid (HI-E), platelet (HI-P), and/or neutrophil (HI-N).
Duration of Response | 24 months
  Duration of response will be measured from the date of initial response until failure (includes death from any cause), relapse (after CR or PR) or progression, as defined by the Modified IWG Response Criteria in MDS.
Event-Free Survival | 24 months
  Duration of event free survival will be measured from the start of treatment until failure (as defined in the Modified IWG Response Criteria) or death from any cause.
Progression-Free Survival | 24 months
  Duration of progression free survival will be measured from the start of treatment until progression (as defined in the Modified IWG Response Criteria) or death from MDS.

IPD SHARING:
Plan to Share IPD: No